CLINICAL TRIAL: NCT03531554
Title: Acute Nutritional Ketosis in VLCAD Deficiency: Testing the Metabolic Base for Therapeutic Use
Brief Title: Acute Nutritional Ketosis in VLCAD Deficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: UMC Utrecht (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); University of Oxford (Other); ESN (Erfelijke Stofwisselingsziekten Nederland) (Unknown)
Responsible Party: Principal Investigator, dr. J.A.L. Jeneson, Principal Investigator, University Medical Center Groningen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: METC2014.492;ABR51222.042.14
Record Dates: First submitted 2017-10-17; First posted 2018-05-21 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: VLCAD Deficiency; Fatty Acid Oxidation Defects
Keywords: Fatty acid Oxidation Disorders; ketone ester; VLCAD deficiency
MeSH Terms: conditions — VLCAD deficiency | interventions — Exercise; Magnetic Resonance Imaging; Positron-Emission Tomography

STUDY DESIGN:
Intervention Model Description: randomized, blinded, placebo controlled, 2-way cross-over trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ketone ester drink (Experimental): Oral intake of ketone ester drink muscle biopsy exercise muscle biopsy Magnetic Resonance imaging
  Interventions: Dietary Supplement: ketone ester drink; Behavioral: exercise; Procedure: muscle biopsy; Diagnostic Test: Magnetic Resonance Imaging
- carbohydrate drink (Placebo Comparator): Oral intake of isocaloric carbohydrate drinkmuscle biopsy exercise muscle biopsy Magnetic Resonance imaging
  Interventions: Behavioral: exercise; Procedure: muscle biopsy; Diagnostic Test: Magnetic Resonance Imaging

INTERVENTIONS:
Dietary Supplement: ketone ester drink — 395 mg of ketone ester/kg
  Other Names: deltaG (R)
  Arms: ketone ester drink
Behavioral: exercise — 35 min cycling test on an upright bicycle, followed by 10 minutes of supine cycling inside a MR scanner.
Procedure: muscle biopsy — biopsy from the quadriceps muscle prior to and immediately after upright bicycling
Diagnostic Test: Magnetic Resonance Imaging — 1H MR images and 31P MR spectra were acquired from the upper leg prior to-, during and after exercise
  Other Names: Magnetic Resonance Spectroscopy

SUMMARY:
To test if a ketone-ester based drink can boost muscle mitochondrial function in vivo in patients with VLCADD in order to establish a rational basis for therapeutic use in this disorder.

DETAILED DESCRIPTION:
Exertional rhabdomyolysis is a common symptom in very long-chain acylCoA dehydrogenase deficient (VLCADD) patients. Failing muscle ATP homeostasis, due to impaired fatty acid oxidation, is the most likely cause. Therefore, supplementation with an alternative energy substrate to boost ATP homeostasis, such as an exogenous ketone ester (KE) drink, could be a therapeutic option. Previous results suggest that KE is preferentially oxidized in the tricyclic acid (TCA) cycle and improves physical endurance in athletes. Our primary objective is to test if KE boosts muscular ATP homeostasis in VLCADD patients to establish a rational basis for therapeutic use.

VLCADD patients will be included in a randomized, blinded, placebo controlled, 2-way cross-over trial. Prior to each test, patients receive a KE drink or an isocaloric carbohydrate equivalent, and completed a 35 min cycling test on an upright bicycle, followed by 10 minutes of supine cycling inside a MR scanner. The protocol will be repeated after at least one week with the opposite drink.

ELIGIBILITY:
Inclusion Criteria:

- Confirmed VLCADD by genetic profiling

Exclusion Criteria:

* contraindications for MRI studies (assessed by standardised questionnaire as previously used in METC 08-267/K; see UMCG section F METC documents)
* inability to perform bicycle exercise.
* recent episode of rhabdomyolysis, or treatment for acute renal failure in the past 2 months.
* intercurrent illness which may influence exercise tolerance (anaemia, musculoskeletal injury, or other undiagnosed illness under investigation).
* known coronary artery disease, positive history for angina, or changes on ECG suggestive of previous ischaemia without a negative stress test.
* insulin-dependent diabetes mellitus.
* loss of, or an inability to give informed consent.
* pregnancy or current breastfeeding, or females not taking the oral contraceptive pill (this is due to the variability in hormonal patterns and substrate levels with different parts of the menstrual cycle).
* any other cause which in the opinion of the investigators, may affect the volunteers ability to participate in the study.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Change of ATP concentration in millimolar | During session 2 and 3: continuous measurements from t=75 minutes until t=85 minutes
  steady-state in vivo intramuscular concentration of ATP metabolites during rest and exercise.
Change of PCr concentration in millimolar | During session 2 and 3: continuous measurements from t=75 minutes until t=85 minutes
  steady-state in vivo intramuscular concentration of ATP metabolites during rest and exercise.
Change of Pi concentration in millimolar | During session 2 and 3: continuous measurements from t=75 minutes until t=85 minutes
  steady-state in vivo intramuscular concentration of ATP metabolites during rest and exercise.

SECONDARY OUTCOMES:
kinetic rate constant of ATP synthesis in Hertz | session 2 and 3, 10 minutes each time
  rate constant of Pi and PCr recovery post-exercise
intramuscular concentration of H+ in millimolar | session 2 and 3, 10 minutes each time
  steady-state in vivo intramuscular concentration of H+ during rest and exercise
completion of 35 minute upright bicycling bout at FATMAX | Session 2 and 3, 35 minutes
  (yes/no; if no, #minutes)
completion of 10 minute supine bicycling bout at FATMAX in scanner | Session 2 and 3, 10 minutes
  (yes/no; if no, #minutes)
HR in beats per minute | During session 1, 15 minutes During Session 2 + 3: 35 minutes
  heart rate, VO2 and VCO2 dynamics. During session 2+3 breath sampling will be done for 2 minutes per timepoint, simultaneously with blood sampling.
VO2 in milliliter per minute per kilogram | During session 1, 15 minutes During Session 2 + 3: 35 minutes
  heart rate, VO2 and VCO2 dynamics. During session 2+3 breath sampling will be done for 2 minutes per timepoint, simultaneously with blood sampling.
VCO2 in milliliter per minute per kilogram | During session 1, 15 minutes During Session 2 + 3: 35 minutes
  VCO2 dynamics during session 2+3 breath sampling for 2 minutes per timepoint, simultaneously with blood sampling.
Changes in blood metabolites: D-betahydroxybutyrate in millimol per liter | Session 2 and 3, 265 minutes per session
  Samples are taken at baseline, 30 minutes, 40 minutes, 50 minutes, 60 minutes, 75 minutes, 85 minutes and 265 minutes after ingestion of the testdrink
Changes in blood metabolites: glucose in millimol per liter | Session 2 and 3, 265 minutes per session
  Samples are taken at baseline, 30 minutes, 40 minutes, 50 minutes, 60 minutes, 75 minutes, 85 minutes and 265 min after ingestion of the testdrink
Changes in blood metabolites: lactate in millimol per liter | Session 2 and 3, 265 minutes per session
  Samples are taken at baseline, 30 minutes, 60 minutes, 85 minutes and 265 min after ingestion of the testdrink
Changes in blood metabolites: insulin in picomol per liter | Session 2 and 3, 265 minutes per session
  Samples are taken at baseline, 30 minutes, 60 minutes, 85 minutes and 265 min after ingestion of the testdrink
Changes in blood metabolites: creatine kinase in units per liter | Session 2 and 3, 265 minutes per session
  Samples are taken at baseline, 30 minutes, 60 minutes, 85 minutes and 265 min after ingestion of the testdrink
Changes in blood metabolites: triglycerides in millimol per liter | Session 2 and 3, 265 minutes per session
  Samples are taken at baseline, 30 minutes, 60 minutes, 85 minutes and 265 min after ingestion of the testdrink
Changes in blood metabolites: LDL cholesterol in millimol per liter | Session 2 and 3, 265 minutes per session
  Samples are taken at baseline, 30 minutes, 60 minutes, 85 minutes and 265 min after ingestion of the testdrink
Changes in blood metabolites: free fatty acids in millimol per liter | Session 2 and 3, 265 minutes per session
  Samples are taken at baseline, 30 minutes, 40 minutes, 50 minutes, 60 minutes, 75 minutes, 85 minutes and 265 min after ingestion of the test drink
Changes in blood metabolites: total cholesterol in millimol per liter | Session 2 and 3, 265 minutes per session
  Samples are taken at baseline, 30 minutes, 60 minutes, 85 minutes and 265 min after ingestion of the testdrink
Changes in blood metabolites: HDL cholesterol in millimol per liter | Session 2 and 3, 265 minutes per session
  Samples are taken at baseline, 30 minutes, 60 minutes, 85 minutes and 265 min after ingestion of the testdrink
Changes in blood metabolites: acylcarnitines in micromol per liter | Session 2 and 3, 265 minutes per session
  Samples are taken at baseline, 30 minutes, 40 minutes, 50 minutes, 60 minutes, 75 minutes, 85 minutes and 265 min after ingestion of the test drink
Subjective exertion | During Session 2 + 3, assessed during blood sampling, 265 minutes per session
  Measured with Borg score (range from 6 (rest) to 20 (extreme exertion)).
height in meters | 1 minute during screening visit
  height of patient
weight in kilogram | 1 minute during screening visit
  weight of patient to dose intervention and normalize outcome parameters
BMI in kg/m^2 | 1 minute during screening visit
  weight and height will be combined to report BMI in kg/m^2
optional: TCA intermediates in muscle tissue (units is ratio of metabolite peak/ internal standard) and will be expressed as fold change from baseline | Session 2+3: before and after exercise, 20 minutes per session
  metabolomics (mass spectrometry) of muscle tissue on a voluntary basis
optional: glycolysis intermediates in muscle tissue (units is ratio of metabolite peak/ internal standard) and will be expressed as fold change from baseline | Session 2+3: before and after exercise, 20 minutes per session
  metabolomics (mass spectrometry) of muscle tissue on a voluntary basis
optional: acylcarnitines in muscle tissue (units is ratio of metabolite peak/ internal standard) and will be expressed as fold change from baseline | Session 2+3: before and after exercise, 20 minutes per session
  metabolomics (mass spectrometry) of muscle tissue on a voluntary basis
optional: D-betahydroxybutyrate in muscle tissue (units is ratio of metabolite peak/ internal standard) and will be expressed as fold change from baseline | Session 2+3: before and after exercise, 20 minutes per session
  metabolomics (mass spectrometry) of muscle tissue on a voluntary basis
optional: capillary density in muscle tissue based on CD31 staining (capillaries per millimeter^2) | Session 2+3: before and after exercise, 20 minutes per session
  individual phenotypic muscle properties on a voluntary basis. Immunohistochemistry.
optional: mitochondrial density based on ATPase, COX-SDH, SDH and NADH staining (intensity per microgram per minute). | Session 2+3: before and after exercise, 20 minutes per session
  individual phenotypic muscle properties on a voluntary basis. Immunohistochemistry.
optional: mitochondrial density based on as citrate synthase activity expressed as absorbance/s/mg. | Session 2+3: before and after exercise, 20 minutes per session
  individual phenotypic muscle properties on a voluntary basis.
optional: parameters for metabolism and mitochondrial function in muscle (AMPK, PPAR gamma, PGC1a, and GLUT4). All expressed as protein content as % of control. | Session 2+3: before and after exercise, 20 minutes per session
  individual phenotypic muscle properties on a voluntary basis. Westernblots.
optional: lipid accumulation based on Oil-Red-O staining (intensity of staining, and percentage positive-stained cells). | Session 2+3: before and after exercise, 20 minutes per session
  individual phenotypic muscle properties on a voluntary basis. Immunohistochemistry.
optional: muscle fiber type composition based on myosin heavy chain profiling. Type I, IIa, IIx fibres will be expressed as % of total fibres. | Session 2+3: before and after exercise, 20 minutes per session
  individual phenotypic muscle properties on a voluntary basis.
optional: muscle fiber type composition based on ATPase staining (intensity/ug/min). Type I, IIa, IIx fibres will be expressed as % of total fibres. | Session 2+3: before and after exercise, 20 minutes per session
  individual phenotypic muscle properties on a voluntary basis. Immunohistochemistry.
optional: glycogen content of muscle based on Periodic acid-Schiff (PAS) staining (intensity per millimeter^2) | Session 2+3: before and after exercise, 20 minutes per session
  individual phenotypic muscle properties on a voluntary basis. Immunohistochemistry.
optional: glycogen content of muscle measured as glucose released after enzymatic digestion with amyloglucosidase expressed as micromol per gram wet muscle weight. | Session 2+3: before and after exercise, 20 minutes per session
  individual phenotypic muscle properties on a voluntary basis.

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen AL Jeneson, PhD, Principal Investigator — Dept of Neuroscience/ Neuroimaging Center Groningen
Locations (2):
- Netherlands (2):
  - Academic Medical Center, Amsterdam, North Holland
  - Dept of Neuroscience/ Neuroimaging Center, Groningen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cox PJ, Kirk T, Ashmore T, Willerton K, Evans R, Smith A, Murray AJ, Stubbs B, West J, McLure SW, King MT, Dodd MS, Holloway C, Neubauer S, Drawer S, Veech RL, Griffin JL, Clarke K. Nutritional Ketosis Alters Fuel Preference and Thereby Endurance Performance in Athletes. Cell Metab. 2016 Aug 9;24(2):256-68. doi: 10.1016/j.cmet.2016.07.010. Epub 2016 Jul 27. PMID 27475046
- [Background] Diekman EF, Visser G, Schmitz JP, Nievelstein RA, de Sain-van der Velden M, Wardrop M, Van der Pol WL, Houten SM, van Riel NA, Takken T, Jeneson JA. Altered Energetics of Exercise Explain Risk of Rhabdomyolysis in Very Long-Chain Acyl-CoA Dehydrogenase Deficiency. PLoS One. 2016 Feb 16;11(2):e0147818. doi: 10.1371/journal.pone.0147818. eCollection 2016. PMID 26881790
- [Derived] Bleeker JC, Visser G, Clarke K, Ferdinandusse S, de Haan FH, Houtkooper RH, IJlst L, Kok IL, Langeveld M, van der Pol WL, de Sain-van der Velden MGM, Sibeijn-Kuiper A, Takken T, Wanders RJA, van Weeghel M, Wijburg FA, van der Woude LH, Wust RCI, Cox PJ, Jeneson JAL. Nutritional ketosis improves exercise metabolism in patients with very long-chain acyl-CoA dehydrogenase deficiency. J Inherit Metab Dis. 2020 Jul;43(4):787-799. doi: 10.1002/jimd.12217. Epub 2020 Feb 5. PMID 31955429

DOCUMENTS (1):
  • Study Protocol (2017-02-15): https://cdn.clinicaltrials.gov/large-docs/54/NCT03531554/Prot_000.pdf